CLINICAL TRIAL: NCT07333742
Title: A Randomized, Open Label, Single Oral Dose, 2x2 Crossover Study to Compare the Pharmacokinetics and Safety/Tolerability of Gemigliptin/Dapagliflozin/Metformin 50/10/1000 mg and Coadministration of Gemigliptin 50 mg and Dapagliflozin/Metformin 10/1000 mg in Healthy Adults in Fed Condition
Brief Title: A Clinical Study to See How the Body Handles and How Safe a Combination Tablet of Gemigliptin, Dapagliflozin, and Metformin 50/10/1000mg is Compared to Taking Gemigliptin 50mg Separately With Dapagliflozin/Metformin 10/1000mg in Healthy Adults After a Meal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LG-GMCL001
Record Dates: First submitted 2025-11-24; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Fed Conditions; Healthy Volunteer
Keywords: Bioequivalence study; Fed condition
MeSH Terms: interventions — Drug Evaluation; LC15-0444; dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Sequence A: Test drug -> Reference drug
  Interventions: Drug: Test drug: Fixed-dose combination (FDC) of gemigliptin/dapagliflozin/metformin 50/10/1000 mg; Drug: Reference drug: gemigliptin (Zemiglo) 50mg, Xigduo XR 10/1000 mg
- Sequence B (Experimental): Sequence B: Reference drug -> Test drug
  Interventions: Drug: Test drug: Fixed-dose combination (FDC) of gemigliptin/dapagliflozin/metformin 50/10/1000 mg; Drug: Reference drug: gemigliptin (Zemiglo) 50mg, Xigduo XR 10/1000 mg

INTERVENTIONS:
Drug: Test drug: Fixed-dose combination (FDC) of gemigliptin/dapagliflozin/metformin 50/10/1000 mg — All participants take 1 tablet of either test drug or reference drug after meal.
Drug: Reference drug: gemigliptin (Zemiglo) 50mg, Xigduo XR 10/1000 mg — All participants take 1 tablet of either test drug or reference drug after meal.

SUMMARY:
Bioequivalence study for the fixed-dose combination of gemigliptin/dapagliflozin/metformin 50/10/1000 mg under fed conditions in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-50 years in healthy volunteers
2. 18.0 kg/m^2 ≤ BMI ≤ 29.9 kg/m^2, 50kg ≤weight ≤ 90kg
3. 60≤ FPG≤125 mg/dL
4. Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial.

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system.
2. Subjects with clinically significant abnormal findings during tests (or examinations)
3. Subjects with a history of hypersensitivity or clinically significant hypersensitivity reactions to test drugs or other drugs
4. Subjects judged ineligible by the investigator

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
The plasma concentration of gemigliptin, dapagliflozin, and metformin | - Period 1: 16 times up to 72 hours from IP administration - Period 2: 16 times up to 72 hours from IP administration
  Primary Parameters: Area under the plasma concentration versus time curve (AUClast) of gemigliptin, dapagliflozin, and metformin
The plasma concentration of gemigliptin, dapagliflozin, and metformin | - Period 1: 16 times up to 72 hours from IP administration - Period 2: 16 times up to 72 hours from IP administration
  Primary Paramenters: Peak Plasma Concentration (Cmax) of gemigliptin, dapagliflozin, and metformin

SECONDARY OUTCOMES:
The plasma concentration of gemigliptin, dapagliflozin and metformin | Period 1: 16 times up to 72 hours from IP administration Period 2: 16 times up to 72 hours from IP administration
  Secondary Parameters: Time to Maximum(Tmax) Concentration of gemigliptin, dapagliflozin, and metformin
The plasma concentration of gemigliptin, dapagliflozin and metformin | - Period 1: 16 times up to 72 hours from IP administration - Period 2: 16 times up to 72 hours from IP administration
  Secondary Parameters: Lag Time(Tlag) of gemigliptin, dapagliflozin, and metformin
The plasma concentration of gemigliptin, dapagliflozin and metformin | - Period 1: 16 times up to 72 hours from IP administration - Period 2: 16 times up to 72 hours from IP administration
  Secondary Parameters: Area Under the Curve to Infinity(AUCinf) of gemigliptin, dapagliflozin, and metformin
The plasma concentration of gemigliptin, dapagliflozin and metformin | - Period 1: 16 times up to 72 hours from IP administration - Period 2: 16 times up to 72 hours from IP administration
  Secondary Parameters: Half-life(t1/2) of gemigliptin, dapagliflozin, and metformin
The plasma concentration of gemigliptin, dapagliflozin and metformin | - Period 1: 16 times up to 72 hours from IP administration - Period 2: 16 times up to 72 hours from IP administration
  Secondary Parameters: Apparent Clearance(CL/F) of gemigliptin, dapagliflozin, and metformin
The plasma concentration of gemigliptin, dapagliflozin and metformin | - Period 1: 16 times up to 72 hours from IP administration - Period 2: 16 times up to 72 hours from IP administration
  Secondary Parameters: Apparent Volume of Distribution(Vz/F) of gemigliptin, dapagliflozin, and metformin

OTHER OUTCOMES:
Assessment - Safety (Adverse events) | up to day 18 (post study visit)
  A list of all adverse events for each treatment group and for all participants with seriousness, severity, relationship with investigational product. A number of participant with adverse event.
Assessment - Safety (Physical examination) | 3 times until 72 hours from IP administration
  Any finding in general condition, nutritional status and other category by medical interview
Assessment - Safety (Vital sign) | 7 times until 72 hours from IP administration
  Systolic Blood Pressure(mmHg), Diastolic Blood Pressure(mmHg), Pulse Rate(beats/min), Temperature(℃)
Assessment - Safety (12-lead ECG results) | 4 times until post-study visit
  Ventricular rate(beats/min), PR interval(msec), QRS(msec), QT(msec), QTcB(msec)
Assessment - Safety (Clinical laboratory test results) | 4 times until post-study visit
  Hematology, Blood Chemistry, Urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No